CLINICAL TRIAL: NCT00116181
Title: A Multicenter, Open-Label, Prospective Study to Evaluate the Effectiveness and Safety of Etanercept in the Treatment of Subjects With Psoriasis-EASE in Psoriasis
Brief Title: Study to Help Understand the Action of the Drug Etanercept for the Adult Patient With Psoriasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Rockefeller University (Other)
Collaborators: Amgen (Industry)
Responsible Party: James Krueger, MD, Rockefeller University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JKR 542
Record Dates: First submitted 2005-06-27; First posted 2005-06-28 (Estimated); Last update posted 2011-03-18 (Estimated); Status verified 2011-03

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — Etanercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- continuous therapy (Experimental): Subjects will receive 50 mg once weekly SC (2 injections of 25 mg etanercept SC within 1 hour once weekly) for weeks 13 through 24.
  Interventions: Drug: Etanercept
- intermittent therapy (Active Comparator): Subjects who achieve a responder status on the PGA (PGA score £ 2 and improved from baseline) at week 12 will discontinue therapy. Upon relapse of PGA responder status, etanercept will be administered 50 mg once weekly SC (2 injections of 25 mg etanercept SC within 1 hour once weekly) through week 24.
  Interventions: Drug: Etanercept

INTERVENTIONS:
Drug: Etanercept — All subjects will administer etanercept 50 mg twice weekly subcutaneously (2 injections of 25 mg etanercept SC within 1 hour twice weekly) for the first 12 weeks of study.
  Subjects randomized to the "continuous therapy" arm will then receive 50 mg once weekly SC (2 injections of 25 mg etanercept SC within 1 hour once weekly) for weeks 13 through 24. Subjects randomized to the "intermittent therapy" arm will be assessed for response. Those who achieve a responder status on the PGA (PGA score £ 2 and improved from baseline) at week 12 will discontinue therapy. Upon relapse of PGA responder status, etanercept will be administered 50 mg once weekly SC (2 injections of 25 mg etanercept SC within 1 hour once weekly) through week 24.

SUMMARY:
The investigator's laboratory is studying a skin disease known as psoriasis. The purpose of this protocol is to study the action and the effects of Etanercept, on psoriasis. This medication has been studied extensively and has been found to be effective and safe in the treatment of psoriasis. The eligible patient will have 10% of his/her body surface area involved with psoriasis vulgaris. This trial is a phase III study to help understand the action of the drug etanercept, trade name Enbrel, for the adult patient with moderate to severe plaque psoriasis and who is a candidate for internal medications.

DETAILED DESCRIPTION:
The eligible patient will receive the drug Etanercept (Enbrel), and will self inject with Etanercept twice a week for the first 12 weeks. The patient will be taught to self inject the medication at home and will be seen in the clinic weekly, for the first four weeks and then once a month.

During the second 12 weeks of the study, patients will be placed in one of two groups by the drug company participating. One group of patients will be randomized to either continue receiving the medication and will self inject once a week. A second group will be randomized to not receive the medication but will continue to be followed and examined at monthly visits. The drug company will do the randomization or choice of group, and each patient has a one in two chance of being placed in one group or the other.

At the clinic visits, the patient can expect that a physical exam and skin exam will be done. At specific weeks, blood work will be drawn, clinical photography taken and a skin biopsy done. Two types of skin biopsies will be done after local anesthesia has been administered. One is a punch biopsy where a small piece of skin will be taken, the approximate size of a pencil eraser. The second type of skin biopsy is a shave biopsy, where a postage sized piece of skin will be taken.

ELIGIBILITY:
Inclusion Criteria:

* Gender: Male and Female
* Minimum Age: 18
* Maximum Age: 70

Exclusion Criteria:

* Healthy Volunteers

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2004-10; Primary Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects achieving a responder status on the Physician's Global Assessment (PGA) at week 24 | screening, baseline, week 2, 4, 12, 16, 20 and 24

SECONDARY OUTCOMES:
Subject incidence rates of serious adverse events, serious infections, non-melanoma skin cancer, and all malignancies | measured over 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: James G. Krueger, MD, PHD, Principal Investigator — Rockefeller University
Locations (1):
- Rockefeller University, New York, New York, United States

REFERENCES:
- See also: Related Info — http://www.rucares.org